CLINICAL TRIAL: NCT04735913
Title: Effects of Metabolic Enzymes and Transporter Gene Polymorphisms on the Pharmacokinetics and Metabolism of Oral Abiraterone Acetate in Healthy Chinese Adults
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Zhongnan Hospital (Other)
Responsible Party: Principal Investigator, Jianying Huang, Principal Investigator, Zhongnan Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 20201010
Record Dates: First submitted 2020-11-16; First posted 2021-02-03 (Actual); Last update posted 2022-01-03 (Actual); Status verified 2021-12

CONDITIONS: Abiraterone Acetate; Gene Polymorphism; Pharmacokinetic; Metabolic Analysis; Plasma Concentration
Keywords: Abiraterone; pharmacokinetic; metabolites; plasma; gene polymorphism
MeSH Terms: interventions — Abiraterone Acetate

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Fasting group (Other): Subjects will take abiraterone acetate tablets (250 mg, produced by Patheon Ich, trade name: Zytiga®) orally on an empty stomach and their blood and plasma samples, urine and faeces samples in 72h will be collected for detection.
  Interventions: Drug: Abiraterone acetate tablets
- Postprandial group (Experimental): Subjects will take abiraterone acetate tablets (250 mg, produced by Patheon Ich, trade name: Zytiga®)orally after meals and their blood and plasma samples, urine and faeces samples in 72h will be collected for detection.
  Interventions: Drug: Abiraterone acetate tablets

INTERVENTIONS:
Drug: Abiraterone acetate tablets — Subjects will take abiraterone acetate tablets (250 mg, produced by Patheon Ich, trade name: Zytiga®) orally on an empty stomach or after meals and their blood and plasma samples, urine and faeces samples in 72h will be collected for detection.

SUMMARY:
1. To explore the relationship between the changes of plasma concentration of abiraterone acetate after taken orally on fasting or postprandial and gene polymorphism.
2. Study of drug Metabolite profiling after oral administration of abiraterone acetate on fasting and postprandial in Chinese adults.

DETAILED DESCRIPTION:
Prostate cancer is the most common malignancy in men currently, second only to lung cancer in China. And in Europe and America, it has already overtaken lung and bowel cancer and become the greatest threat of of men's health. After the diagnosis of high-risk prostate cancer patients, endocrine therapy is still the main treatment. It is effective for most patients who receive androgen deprivation therapy at first. However, after the remission whose median time is 18 to 24 months through endocrine therapy, most patients will turn to castration resistant prostate cancer (CRPC). The treatment of CRPC has always been a difficult point , and now it has become the emphasis of new endocrine drug development for prostate cancer.

Abiraterone acetate tablets in combination with prednisone apply to the treatment of metastatic castration-resistant prostate cancer. It has been approved by the US Food and Drug Administration in 2011 and gotten listing license in China. Abiraterone acetate is an effective irreversible inhibitor CYP17 enzyme and can be converted into abiraterone in vivo. Abiraterone is an androgen biosynthesis inhibitor with a high affinity and selectivity to CYP17. The inhibitory activity of abiraterone for CYP17 was 10-30 times higher than that of ketoconazole. Androgen biosynthesis is inhibited by inhibiting CYP17. The results of many large-scale clinical trials showed that abiraterone acetate could effectively prolong survival time of the patients .

In this study, Blood and plasma samples, urine and faeces samples in 72h from healthy Chinese adult volunteers who have taken abiraterone acetate tablet orally on an empty stomach or after meals were collected for metabolite analysis, the relationship between plasma concentration and gene polymorphism, and identifying the major metabolites in metabolic biological samples to reveal the pharmacokinetic characteristics of abiraterone acetate tablets，demonstrate the pharmacodynamic mechanism，and explore the effect of different genotypes Pharmacokinetic characteristics in healthy Chinese adults.

The result provides theoretical basis for clinical rational drug use.

ELIGIBILITY:
Inclusion Criteria:

* Age: Healthy male subjects aged 18 to 65 years
* Weight: weight ≥50.0kg, 19 ≤ BMI ≤ 26 kg/m2, BMI=weight (kg) / height2(m2)
* Fully aware of the purpose, nature, method and possible adverse reactions of the study, and sign informed consent prior to the commencement of any study procedure on a voluntarily base.
* Be able to communicate well with the investigator and understand and abide by the terms of the study requirements.

Exclusion Criteria:

* Clinical laboratory examination is abnormal and clinically significant.
* Vital signs examination is abnormal and clinically significant, or there are other diseases of clinical significance（Including but not limited to gastrointestinal tract, kidney, liver, nerve, blood, endocrine, tumor, lung, immune, mental or cardio-cerebrovascular disease）or other specific systemic disease.
* Electrocardiogram is abnormal and clinically significant.
* HbsAg, Anti - HCV, TPPA, or HIV antibody positive.
* History of allergy to abiraterone acetate tablets or its ingredients and analogs
* The number of daily smoking >5 during 3 months before the trial.
* Alcoholics or regular drinkers in the 6 months prior to the trial, that is drinking more than 14 units per week (1 Unit =360mL beer or 45mL 40% liquor or 150mL wine)
* Positive for drug, has a history of drug abuse in the past five years or has used drugs in the 3 months prior to the trial.
* Positive for alcohol screening or use of any alcoholic product within 24 hours prior to taking the study drug.
* Blood donation or massive blood loss within 3 months prior to taking the study drug (>450mL).
* Take any xanthine rich beverage, food, grapefruit fruit or products that contain grapefruit in 48 hours before the trial.
* Take in chocolate or any food or drink containing caffeine in 48 hours before the trial.
* A history of dysphagia or any gastrointestinal disease that affect drug absorption.
* Have taken the study drug or participated in the drug or medical device within three months before this trial.
* There are major changes in diet or exercise habits recently.
* Acute disease occurs during the study screening phase or prior to taking study drugs.
* There are drug combination of CYP3A4, P-GP, or Bcrp inhibitors or inducers (such as itraconazole, ketoconazole, dronedarone et al.), or any drugs that affect hepatic microsomal enzyme activity during the 28 days before taking the study drug.
* Accompanied by any coagulation disorders (such as Willebrand's disease or hemophilia) or history of hemorrhagic disease.
* Accompanied by any disease that increases the risk of bleeding, such as hemorrhoids, acute gastritis, stomach or duodenal ulcers, etc.
* Special requirements on diet and fails to comply with the diet provided and the corresponding regulations, especially for the lactose intolerant.
* History of asthma or seizures.
* Have a pregnancy plan in 6 months, sperm or egg donation, or reluctance to use one or more non-drug contraceptives during the trial.
* Taking any prescription drugs, nonprescription drug, over-the-counter, vitamin products, or herbal medicines in 14 days before taking the study drug.
* Patients with abnormal nucleic acid or antibody detection of COVID-19 and considered ineligible by the investigator.
* Pulmonary CT were abnormal and considered inappropriate to participate in the study by the investigator.
* Subjects considered to have poor compliance or have any factors that would make them inappropriate to participate in the study.

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 81 (Estimated)
Dates: Start 2020-05-05 (Actual); Primary Completion 2020-08-20 (Actual); Study Completion 2022-07-01 (Estimated)

PRIMARY OUTCOMES:
Concentrations of abiraterone in plasma | 2 months
  -1h, 30min, 1h , 1.5h, 2h, 2.5h, 3h, 4h, 5h, 6h, 8h, 12h, 24h, 36h, 48h, 60h, 72h after administration for blood sampling
Cmax | 2 months
  peak concentration
AUC0-t | 2 months
  Area under curve. The linear trapezoid method is used to calculate the blood drug concentration from zero to the last measurable concentration area under the curve
AUC0-∞ | 2 months
  The area under the blood concentration-time curve from zero to infinite blood concentration
λz | 2 months
  End phase elimination rate constant, the least square method is used to find the slope of the optimal curve for phase elimination And multiplied by 2.303
T1/2z | 2 months
  Elimination or final half-life, 0.693/λz
AUC_%Extra | 2 months
  [（AUC0-∞- AUC0-t）/ AUC0-∞]×100%, Percentage of residual area
Vz/F | 2 months
  apparent volume of distribution, Vz/F = CLz/F /λz
CLz/F | 2 months
  apparent clearance, CLZ /F= administration dose /AUC0-∞
the main metabolite of abiraterone | 2 months
  The plasma, urine and feces samples were collected to assay the metabolic profile of abiraterone in vivo by UFLC-Q-Exactive Orbitrap HRMS system
genotyping related to abiraterone metabolism | 10 months
  Mutation sites of transporter and metabolic enzyme related to abiraterone metabolism were detected through the gene detection technology service platform

CONTACTS AND LOCATIONS:
Locations (1):
- Zhongnan Hospital of Wuhan University, Wuhan, Hubei, China